CLINICAL TRIAL: NCT07312279
Title: Study on the Efficacy of Temporal Interference Stimulation (TIS) for Parkinson's Disease
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zhongnan Hospital (Other)
Responsible Party: Principal Investigator, BinMei, Attending Physician, Zhongnan Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025267
Record Dates: First submitted 2025-12-12; First posted 2025-12-31 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Temporal Interference Stimulation (TIS); Parkinson's Disease
Keywords: TIS; Parkinson; UPDRS
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- A:STN (Experimental): The subthalamic nucleus (STN) stimulation target
  Interventions: Device: TIS

INTERVENTIONS:
Device: TIS — Temporal Interference Stimulation

SUMMARY:
The primary objective of this clinical study is to evaluate the therapeutic efficacy of Temporal Interference Stimulation (TIS), a non-invasive deep brain stimulation technique, in patients with Parkinson's disease, and to further investigate its potential mechanisms of action. Although TIS offers lower stimulation intensity and precision compared to conventional Deep Brain Stimulation (DBS), it possesses the distinct advantage of being non-invasive. This study utilizes TIS to explore different stimulation targets analogous to those used in DBS for Parkinson's disease, thereby providing valuable insights for subsequent DBS surgical interventions. The findings will contribute preliminary exploratory evidence regarding the application of non-invasive deep brain stimulation technology in the treatment of Parkinson's disease.

ELIGIBILITY:
Inclusion Criteria:

1. Adult males or females aged 40 years or above;
2. Diagnosed with idiopathic Parkinson's disease according to the UK Brain Bank Criteria, with onset after 40 years of age;
3. Previous or current dopaminergic replacement therapy (e.g., levodopa) with good response; (4) Hoehn and Yahr (H&Y) stage 1.5-2.5;
4. Ability to walk independently without assistive devices for at least 5 minutes;
5. Absence of severe freezing of gait (FOG);
6. Disease duration ≥2 years since diagnosis, with stable clinical condition and ability to comply with study assessments and interventions;
7. Stable medication dosage for at least 4 weeks prior to the study;
8. Hoehn and Yahr (H&Y) stage 1.5-2.5;
9. Signed informed consent, with the participant or legal guardian capable of understanding and willing to participate in the study.

Exclusion Criteria:

1. Presence of other neurological disorders that may interfere with the study
2. Mild or greater cognitive impairment (MoCA score ≤23)
3. Orthopedic or other health conditions that may affect gait or balance
4. Contraindications to MRI scanning, such as claustrophobia
5. History of antipsychotic, antidepressant, or other medications that may affect dopamine levels
6. Other significant psychiatric history
7. Contraindications including history of epilepsy, traumatic brain injury, or implanted metal devices in the brain or heart (e.g., stimulators, pacemakers)
8. History of electroconvulsive therapy
9. Concurrent participation in other gait- or balance-related intervention training
10. Physician-diagnosed cardiovascular risk factors for exercise.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-12-30 (Estimated); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
UPDRS-3 | From enrollment through the 3-month follow-up
  Changes in the Movement Disorder Society-Unified Parkinson's Disease Rating Scale Part III (MDS-UPDRS III) scores from baseline to immediately after and 1 month after a single treatment session.

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2025-09-04): https://cdn.clinicaltrials.gov/large-docs/79/NCT07312279/Prot_SAP_ICF_000.pdf